CLINICAL TRIAL: NCT03208686
Title: Self-Management of Diabetes in Black Men
Brief Title: The Men Are Now United Program
Acronym: MANUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other); Claremont Graduate University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CGA#149084
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Type2 Diabetes
Keywords: Gender; Men; Black/African American; Self-management
MeSH Terms: conditions — Coitus; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Other): A single-arm intervention comprised of discussion groups, text messages, and a cloud-based cellular glucometer.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — A single-arm intervention comprised of (a) 10 weekly discussion groups; (b) motivational text messages; (c) a remote sensing persuasive health technology - a cloud-based cellular glucometer connected to a dedicated web site to reduce A1c by 0.5% by improving diabetes self-management behaviors.

SUMMARY:
The purpose of this application is to create and implement a targeted, culturally grounded, diabetes self-management intervention for Black men that uses social support, mobile health, and remote sensing technology to improve diabetes-related outcomes.

DETAILED DESCRIPTION:
The investigators propose a single-subject, repeated measures intervention where each participant will serve their own control. Participants will serve as their own controls for a period of three months prior to the start of the four-month intervention. The study will conclude with an assessment 7-months from baseline. Single-subject designs are most often used in applied research. The design allows the participant to serve as the control, rather than using another individual/group. The design is sensitive to individual differences whereas group designs are sensitive to averages of groups. Year 1 is dedicated to the development of the text messages and the content for the 10 group meeting sessions. Year 2 focuses on the Time-1 control period assessment (pre-baseline at 3 months before the intervention), the Time-2 assessment (baseline), implementation of the 10-week intervention, a post-intervention assessment (Time-3), and 3-month follow up at Time-4, and analysis. Specifically, in Year 2, the primary outcome of A1c will be assessed at Time-1, 3 months later at the start of the intervention, at the end of the intervention, and at 7-months. The investigators will also include secondary assessments of glucose readings, waist circumference, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Black/African American
* Male
* Tyep 2 Diabetes
* 21 years old or older
* Owns cell or smart (mobile) phone or willing to use one if provided

Exclusion Criteria:

* Non-ambulatory
* Serious physical illness
* Psychiatric diagnosis of serious mental illness
* Serious diabetes complications impeding meaningful participation

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification
Enrollment: 41 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | 4 Months
  A1c

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, Flint, Michigan, United States